CLINICAL TRIAL: NCT01679158
Title: Evaluating MOTIlity, Hormonal Impact, Satiety, and Weight Changes With VArying Procedural TEchniques Utilizing the Incisionless Operating Platform for the Treatment of Primary Obesity
Brief Title: MOTIVATE Weight Loss Study
Acronym: MOTIVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USGI Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPR600
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: Using POSE as a treatment for Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Continuous Horizontal row (Experimental): Use the IOP system from USGI to install suture anchors running from the distal body into the proximal antrum
  Interventions: Device: Using The IOP system from USGI to place suture anchors
- Reduction in "ring" opening (Experimental): Use the IOP system from USGI to install suture anchors to reduce the "ring" opening to the antrum
  Interventions: Device: Using The IOP system from USGI to place suture anchors
- Control Arm (Experimental): Use the IOP system from USGI to install suture anchors in the Current V shape in distal body
  Interventions: Device: Using The IOP system from USGI to place suture anchors

INTERVENTIONS:
Device: Using The IOP system from USGI to place suture anchors — Sutures are placed in the distal body in one of three randomized techniques:
  "A" = reduction in "ring" opening to antrum using plications "B" = continuous horizontal row, running from distal body into proximal antrum "C" = Control. Current V shape as Control
  Other Names: The g-Cath EZ Suture Anchor Delivery Catheter

SUMMARY:
The purpose of this study is to evaluate the impact of minor variations in Incisionless Operating Platform (IOP)procedural techniques on gastric emptying, hormone levels, satiety, and weight loss in the treatment of primary obesity. It will confirm, in an open prospective study, the action mechanisms for the "POSE" endoscopic treatment technique for obesity, and it will help determine if they are maintained at least 6 months following the procedure. Durability of weight loss will be tracked through post-POSE visits up to 18 months following the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Has a BMI of >30 and <40
2. Male or female ≥21 yrs. of age and < 60 yrs. of age at time of enrollment
3. Patient has had no significant weight change (+/- 5% of total body weight) in last 6 months but has been able to lose significant weight in the past with diet and exercise.
4. Is a reasonable candidate for general anesthesia
5. Agrees not to have any additional weight loss interventional procedures or liposuction for at least 18 months following study enrollment and agrees not to take any prescription or over the counter weight loss medications for at least 1 year.
6. Physically and mentally able to comply with the visit schedule, ancillary testing, and behavior modification (diet and exercise) required for the study and agrees to study commitment requirements
7. Had successful completion of the pre-screening, nutritional and educational programs and psychological assessment supporting that the subject is an appropriate bariatric surgical candidate

Exclusion Criteria:

1. History of (or intra-operative evidence of) bariatric, gastric or esophageal surgery
2. Esophageal stricture or other anatomy and/or condition that could preclude passage of endoluminal instruments
3. Moderate to severe Gastro-esophageal reflux disease (GERD)
4. Known hiatal hernia >3cm by history or as determined by UGI exam or endoscopy
5. Known GI motility disorder or pancreatic insufficiency/disease
6. Intra-operative Exclusion: Active peptic ulcer or hiatal hernia >3cm
7. Pregnancy.
8. Present Corticosteroid Use
9. History of inflammatory disease of GI tract
10. Severe coagulopathies, hepatic insufficiency or cirrhosis
11. History or present use of insulin or insulin derivatives for treatment of diabetes
12. Had Type II Diabetes Mellitus (as defined by HgbA1c >6.0) for greater than 2 years at the time of enrollment
13. Uncontrolled Type II DM (HgbA1c >7.0 at screening)
14. Patient has quit smoking within last 6 months at time of enrollment or plans to quit smoking in the next year
15. Patient has a history of drug or alcohol abuse or actively abusing either
16. Patient is presently being treated with medication for depression, psychosis, or other mood or eating disorder
17. Non-ambulatory or has significant impairment of mobility
18. Works for, or is first degree relative of investigator, study institution, or support staff involved in the study.
19. Known hormonal or genetic cause for obesity
20. Participating in another clinical study
21. Patient is on medications known to impact GI motility or gut hormones that cannot be discontinued prior to nuclear testing
22. Have work hours, family obligations or transportation issues that could interfere with patient returning for all scheduled evaluations, tests and nutritional counseling.
23. Lives >60 kilometers from investigator site.
24. Patient is not able to provide written informed consent

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Weight Loss | Monthly post procedure out to 18 months
  Each patient's weight will be measured and recorded on a monthly basis out to 18 months post procedure

SECONDARY OUTCOMES:
Fasting/Post-prandial Peptides | pre-procedure & 8 weeks post procedure
  1. Samples to be collected when fasting and 30, 60, 90, and 120 minutes after a standard meal (a meal consisting of 400 calories), The meal must be consumed within 10 minutes.. Serum collection tubes will be centrifuged immediately at 4°C for 10 minutes at 3600rpm and stored at -20°C
  2. Samples to be collected by ELISA are: C-peptide, serum insulin, glucose, PYY, GLP-1 (active), leptin, and GIP. Total ghrelin level to be analyzed by RIA.

OTHER OUTCOMES:
Gastric Emptying | Pre-procedure & 2 & 6 months post procedure
  This test consists of determining the duration of a radioactive marker in a stomach, which is non-absorbable, and free of any food components.
Satiety Testing | Pre-procedure & 2 & 6 months post procedure
  The subjects ingest a nutritional drink (Ensure) at a constant rate of 30 mL per minute, constantly filling the glass with a perfusion pump (Gemini PC-2, IMED, San Diego, CA). (The subjects are not conscious of the volume being ingested.) The subjects are instructed to maintain consumption at the fill rate. Participants take note of their sensation of satiety with a graphical classification scale, which combines verbal descriptors on a scale of 0 to 5 (0 = no symptoms, 1 = first sensation of fullness [threshold]; 2 = light, 3 = moderate, 4 = severe, and 5 = maximum fullness or unbearable). The participants are told to stop taking the food product when a score of 5 is obtained. The maximum consumption of volume of the nutritional drink is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge C. Espinos, MD, Principal Investigator — Centro Medico Teknon
Locations (1):
- Centro Medico, Barcelona, Catalonia, Spain